CLINICAL TRIAL: NCT02750839
Title: Influence of Osteoporosis on Clinical Outcomes of Mini-invasive Surgical Treatment of Proximal Humerus Fractures
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Azienda Ospedaliera Bolognini di Seriate Bergamo (Other)
Responsible Party: Principal Investigator, Riccardo Compagnoni, Medical doctor, Azienda Ospedaliera Bolognini di Seriate Bergamo
Other Study IDs: Trevisan
Record Dates: First submitted 2016-04-19; First posted 2016-04-26 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Osteoporosis; Humerus Fracture
MeSH Terms: conditions — Osteoporosis; Humeral Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- proximal humerus fracture: Patients with proximal humerus fracture treated with mini-invasive plate.
  Interventions: Procedure: proximal humerus fracture fixation

INTERVENTIONS:
Procedure: proximal humerus fracture fixation — Mini-invasive proximal humerus fixation with plate, patient in beach chair position, general anesthesia, a small incision lateral to shoulder is made to insert the plate under scope control

SUMMARY:
Aim of the study is to analyze results of treatment of proximal humerus fractures with mini-invasive technique and plate fixation.

In all the patients a analysis of presence of osteoporosis will be done, clinical and x-ray results will be statistically analyzed to evidence any connection between clinical outcomes and osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Proximal humerus fracture

Exclusion Criteria:

* High risk to surgery (ASA 4 - 5)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with proximal humerus fracture, treated with a mini-invasive technique plate.
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2016-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
correlate osteoporosis (Cortical index) with clinical (Constant score) and radiological (X-ray) results of the procedure | 30 months average
  Osteoporosis will be analyzed with the cortical Index, already described in previous articles about this topic. Clinical evaluation will consider the Constant score, the most used functional score for shoulder. X-ray evaluation will analyze the healing of the fracture, studied by a radiologist, and mobilization of the plate or screws. Data will be combined to analyze correlation between clinical results, plate and screws stability and osteoporosis.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Trevisan, Chief, Study Chair — Azienda Ospedaliera Bolognini di Seriate Bergamo

IPD SHARING:
Plan to Share IPD: Undecided